CLINICAL TRIAL: NCT03142477
Title: Effects of Therapeutic Touch in Patients With Female Genital Neoplasia: a Randomized Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Rubens Lene Carvalho Tavares, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 52649715.9.0000.5149
Record Dates: First submitted 2017-05-02; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Quality of Life; Gynecologic Neoplasm; Gynecologic Cancer; Palliative Care; Therapeutic Touch; Reiki
Keywords: Therapeutic touch; Reiki; Laying-on-of-Hands; Spiritual Therapies
MeSH Terms: conditions — Genital Neoplasms, Female | interventions — Surveys and Questionnaires; Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into tree different groups: control, placebo, treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other): Control group patients will not receive any interventions with therapeutic touch. Two different quality of life questionnaires (WHOQOL-Bref and EORTC QLQ-C30) will be applied before and after treatment. Levels of cortisol, salivary IgA, hematological index results and telomerase activity before and after the use of therapeutic touch will be measured.
  Interventions: Other: Questionnaires
- Placebo (Placebo Comparator): Placebo patients group patients will receive the therapeutic touch intervention by a graduate student without any therapeutic touch training. Two different quality of life questionnaires (WHOQOL-Bref and EORTC QLQ-C30) will be applied before and after treatment. Levels of cortisol, salivary IgA, hematological index results and telomerase activity before and after the use of therapeutic touch will be measured.
  Interventions: Other: Questionnaires; Other: Placebo therapeutic touch
- Treatment (Experimental): Treatment patients group patients will receive the therapeutic touch interventions with a trained therapeutic touch professional. Two different quality of life questionnaires (WHOQOL-Bref and EORTC QLQ-C30) will be applied before and after treatment. Levels of cortisol, salivary IgA, hematological index results and telomerase activity before and after the use of therapeutic touch will be measured.
  Interventions: Other: Questionnaires; Other: Therapeutic touch

INTERVENTIONS:
Other: Questionnaires — Two different quality of life questionnaires (WHOQOL-Bref and EORTC QLQ-C30) will be applied before and after treatment. No true or placebo therapeutic touch intervention will be performed.
Other: Placebo therapeutic touch — Placebo therapeutic touch will be done by graduate students without any specific training. The students are instructed to perform the placebo therapeutic touch with no objective intention of improving the patient's health.
  Arms: Placebo
Other: Therapeutic touch — Therapeutic touch will be done by therapeutic touch trained professionals graduate students without any specific training with the intention of improving the patient's health.
  Arms: Treatment

SUMMARY:
This is a randomized controlled prospective study on the use of therapeutic touch in patients diagnosed with gynecological cancer. The patients will be randomized into three groups: control group (will not receive any interventions with therapeutic touch), placebo group (will receive simulated therapeutic touch intervention by individual not knowing this technique) and treatment group(will receive therapeutic touch intervention by a trained therapeutic touch therapist). Two different quality of life questionnaires will be applied (before and after treatment). Levels of cortisol, salivary IgA, hematological indices and telomerase activity before and after the use of therapeutic touch will be compared between groups.

DETAILED DESCRIPTION:
This project is a randomized controlled prospective study on the use of therapeutic touch in patients diagnosed with gynecological cancer. The patients will be randomized into three groups: control group (will not receive any interventions with therapeutic touch), placebo group (will receive simulated therapeutic touch intervention by individual not knowing the practice) and treatment group (will receive therapeutic touch intervention by a trained therapeutic touch therapist). Two different quality of life questionnaires (World Health Organization quality of life questionnaire - WHOQOL-Bref and the quality of life Core-30 questionnaire - EORTC QLQ-C30) from the European Organization for Research and Treatment of Cancer will be applied before and after treatment. Levels of cortisol, salivary IgA, hematological indices and telomerase activity before and after the use of therapeutic touch will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* age over 18 years
* diagnosis of neoplasms of the female genitalia
* Signature of the consent form

Exclusion Criteria:

* history of previous contact with the therapeutic touch technique
* use of psychotropic drugs, severe neurological or psychiatric disorders that make it impossible to participate in the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — eligibility is based on self-representation
Enrollment: 90 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life | up to 16 weeks of follow-up
  Quality of life questionnaire WHOQOL-Bref

SECONDARY OUTCOMES:
Salivary cortisol | Between 10 to 16 weeks
  Salivary cortisol will be measured after the use of therapeutic touch
Quality of life 2 | up to 16 weeks of follow-up
  Quality of life questionnaire EORTC QLQ-C30
Telomerase activity | up to 16 weeks of follow-up
  Telomerase activity will be measured after the use of therapeutic touch

CONTACTS AND LOCATIONS:
Overall Officials: Rubens Tavares, MD, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No